CLINICAL TRIAL: NCT02010086
Title: Cognitive Behavioral Therapy for Core Autism Symptoms in School-Age Children
Brief Title: Schema, Emotion and Behavior-Based Therapy for School Children
Acronym: SEBASTIEN JR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jeffrey J. Wood, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12000556; Autism Speaks 7552 (Other Grant/Funding Number: Autism Speaks 7552)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Intervention; Autism; Treatment sensitivity; School aged; Cognitive behavioral therapy; Social Skills Intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Individual Cognitive Behavioral Therapy
- Standard Community Treatment (Active Comparator)
  Interventions: Behavioral: Standard Community Treatment

INTERVENTIONS:
Behavioral: Individual Cognitive Behavioral Therapy — Therapists will work with families for 32 weekly sessions, each lasting 90 minutes, implementing the CBT manual for children with ASD (Wood et al., 2007).
  Arms: Individual Cognitive Behavioral Therapy
Behavioral: Standard Community Treatment — In this condition, the child meets with a therapist for 32 weekly sessions, each 90 minutes. Therapists use an established manual to provide a standard community therapy treatment.
  Arms: Standard Community Treatment

SUMMARY:
The study is a randomized controlled trial to examine the efficacy of individual cognitive behavioral therapy (CBT) relative to a standard community treatment, in youngsters with autism spectrum disorder (ASD). The individual CBT program has been tailored over the last five years to the clinical needs of high-functioning youth with ASD.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is among the most common childhood developmental disorders. A key goal in the field is the discovery of methods that reduce core autism symptoms. Core autism symptoms include social-cognitive impairments, pragmatic language deficits, and repetitive and rigid behaviors. The core symptoms tend to be stable and resistant to intervention. Most treatments involve group-based social skills training (SST), with limited effects. No treatment for core autism symptoms in school-aged children with ASD meets American Psychological Association guidelines for possible efficacy. Cognitive behavioral therapy (CBT) offers a novel approach for addressing core autism symptoms in higher functioning school-age youngsters. Initial results suggest that individual CBT may also be promising for reducing core autism symptoms (Wood et al., 2009b; Drahota, Wood et al., 2011). The treatment is based on a contemporary model of memory retrieval competition, employing strategies for enhancing the retention of adaptive conceptual and behavioral responses and the suppression of idiosyncratic beliefs and behaviors in daily social contexts, emphasizing the use of deep semantic processing to enhance memory retrieval. We are proposing a randomized controlled trial to examine the efficacy of individual CBT relative to a standard community treatment for youngsters with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Meets research criteria for a diagnosis of autism, based on child scores on the ADI-R and ADOS tests.
* If taking medication, have maintained a stable dose for 1 month prior to baseline assessment.
* Between the ages of 6-9 years.
* The child's teacher consents to participate in the study to play a modest role in helping implement the intervention and facilitate the school observation assessment.

Exclusion Criteria:

* IQ less than 85.
* The child starts taking new medication(s) or current medication dose changes either (a) less than 1 month prior to the diagnostic evaluation, or (b) during the study period.
* The child is participating in an intensive early intervention program for autism such as applied behavior analysis or floortime.
* For any reason the child or parents appear unable to participate in the treatment program.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2011-12 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Playground Observation of Peer Engagement scale | Post-Treatment (week 32)
  An independent evaluator-rated school playground observational measure of joint engagement, which is a valid measure of core autism symptoms with established treatment sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Jeffrey Wood, Los Angeles, California, United States

REFERENCES:
- [Derived] Wood JJ, Kuhfeld M, Sturm A, Cai L, Wood KS, Cornejo Guevara MV, Galan CA, Johnson AR, Cho AC, Weisz JR. Personalized autism symptom assessment with the Youth Top Problems Scale: Observational and parent-report formats for clinical trials applications. Psychol Assess. 2022 Jan;34(1):43-57. doi: 10.1037/pas0001065. Epub 2021 Aug 30. PMID 34460285
- [Derived] Wood JJ, Sze Wood K, Chuen Cho A, Rosenau KA, Cornejo Guevara M, Galan C, Bazzano A, Zeldin AS, Hellemann G. Modular cognitive behavioral therapy for autism-related symptoms in children: A randomized controlled trial. J Consult Clin Psychol. 2021 Feb;89(2):110-125. doi: 10.1037/ccp0000621. PMID 33705167